CLINICAL TRIAL: NCT07200362
Title: A Prospective Cohort Study of Compound Nanxing Zhitong Ointment in the Treatment of Chronic Pain in the Musculoskeletal System
Brief Title: Study of Compound Nanxing Zhitong Ointment in the Treatment of Chronic Pain in Musculoskeletal System
Status: Completed | Type: Observational
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CYZZ2038026 SU
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Primary Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: Use Compound Nanying zhitong Ointment alone, or use it in conjunction with conventional Western medicine treatment, without using any other similar Chinese patent medicines or traditional Chinese medicines.
  Interventions: Drug: Compound Nanying zhitong Ointment
- The non-exposure group: Do not use any other similar proprietary medicines or traditional Chinese medicines.
  Interventions: Other: Do not use any other similar proprietary medicines or traditional Chinese medicines.

INTERVENTIONS:
Drug: Compound Nanying zhitong Ointment — Use Compound Nanying Pain Relief Ointment alone, or use it in conjunction with conventional Western medicine treatment, without using any other similar Chinese patent medicines or traditional Chinese medicines.
  Groups: exposed group
Other: Do not use any other similar proprietary medicines or traditional Chinese medicines. — Do not use any other similar proprietary medicines or traditional Chinese medicines.
  Groups: The non-exposure group

SUMMARY:
A prospective cohort study on the treatment of chronic pain in the musculoskeletal system with Compound Nanxing Pain Relief Ointment. This study adopted an observational research design. Through a cohort study, patient medical records were collected to meet the criteria of chronic pain classification in International Classification of Diseases 11th Revision (ICD-11), which is located in the musculoskeletal system and occurs in the neck and shoulders, waist and back, limbs, and meets the diagnostic criteria of "cold syndrome" in traditional Chinese medicine. The target population was selected to evaluate the clinical effects of Compound Nanxing Pain Relief Ointment in treating chronic pain in the musculoskeletal system, reducing pain, improving muscle and bone function status, and enhancing quality of life. The study aimed to compare the heterogeneity of the clinical effects of Compound Nanxing Pain Relief Ointment in treating chronic pain in the musculoskeletal system. The study plan included 3000 patients, and no intervention in treatment and medication was provided to the patients during the observation period. The shortest medication duration was 2 weeks, and the longest observation period was 3 months.

ELIGIBILITY:
Inclusion Criteria:

For those who visit the orthopedics department, rheumatology department, or pain clinic:

1. Those whose pain is located in the musculoskeletal system as classified in International Classification of Diseases 11th Revision(ICD-11) for chronic pain, and occurs in the neck, shoulders, waist, back, or limbs;
2. Those who meet the diagnostic criteria of "cold syndrome" in traditional Chinese medicine, and their chronic pain worsens or occurs when exposed to cold;
3. Those with continuous or intermittent pain lasting more than 3 months, and without surgical indications.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For those who visit the orthopedics department, rheumatology department, or pain clinic:
  1. Those whose pain is located in the musculoskeletal system as classified in International Classification of Diseases 11th Revision(ICD-11) for chronic pain, and occurs in the neck, shoulders, waist, back, or limbs;
  2. Those who meet the diagnostic criteria of "cold syndrome" in traditional Chinese medicine, and their chronic pain worsens or occurs when exposed to cold;
  3. Those with continuous or intermittent pain lasting more than 3 months, and without surgical indications.
Sampling Method: Non-Probability Sample
Enrollment: 3029 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Global Pain Assessment Scale score | The scores of the Global Pain Assessment Scale were evaluated on Day1, as well as at the 2nd, 4th, 8th, and 12th weeks after the treatment.
  There are a total of 20 items, each rated on a scale of 0 to 10. The total score is calculated by adding up the scores of all items and then dividing by 2. The score range is from 0 to 100. The higher the score, the more severe the pain and its impact.

SECONDARY OUTCOMES:
Pain relief time | The scores of the Global Pain Assessment Scale were evaluated on Day1, as well as at the 2nd, 4th, 8th, and 12th weeks after the treatment.
  The time required for the VAS score to decrease by ≥50% compared to the baseline.The shorter the duration of pain relief, the better the therapeutic effect.
Time when pain disappears | The scores of the Global Pain Assessment Scale were evaluated on Day1, as well as at the 2nd, 4th, 8th, and 12th weeks after the treatment.
  The time required for the pain VAS score to be ≤ 2 points and to remain at that level for 24 hours or more.
Number of days without pain episodes | The scores of the Global Pain Assessment Scale were evaluated on Day1, as well as at the 2nd, 4th, 8th, and 12th weeks after the treatment.
  Record the number of days each month when the patient's affected area is free from pain.
Score of TCM syndromes/signs | The TCM syndrome scores were evaluated on Day 1, as well as at the 2nd, 4th, 8th, and 12th weeks after the treatment.
Score of the Short Form 12 Health Survey (SF-12) | The Short Form 12 Health Survey (SF-12) test was evaluated on day1, as well as at the 2nd, 4th, 8th and 12th weeks after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China